CLINICAL TRIAL: NCT05706909
Title: The Use of Genex in the Management of Early-Stage Osteonecrosis of the Femoral Head
Acronym: Genex
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Biocomposites Ltd (Industry)
Responsible Party: Principal Investigator, Nicolas Piuzzi, Nicolas Piuzzi, M.D., The Cleveland Clinic
Other Study IDs: 22-580
Record Dates: First submitted 2023-01-06; First posted 2023-01-31 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Avascular Necrosis; Osteonecrosis
Keywords: avascular necrosis; osteonecorsis; hip; femoral head
MeSH Terms: conditions — Osteonecrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Genex with ABMC: Injection of autologous bone marrow concentrate and the use of genex® Bone graft Substitute as an adjunct associated with the Core decompression procedure
  Interventions: Device: Genex with ABMC

INTERVENTIONS:
Device: Genex with ABMC — Core decompression, injection of autologous bone marrow concentrate and the use of genex® Bone graft Substitute as an adjunct associated with the decompression procedure

SUMMARY:
The purpose of this study is to assess the clinical and x-ray results of patients who are treated with core decompression of the hip and the injection of a bone marrow concentrate and the use of the Bone Graft Substitute Genex®.

DETAILED DESCRIPTION:
Avascular necrosis (AVN) or osteonecrosis (ON) of the femoral head refers to a condition in bone metabolism when cells of the trabecular bone (porous bone found at the end of long bones like the femur) in the hip spontaneously die. Depending on the amount of femoral head involvement, parts of the surface, like the articular surface that do not have blood vessels may collapse as the disease advances. Although the exact common occurrence of AVN or ON is unknown, the incidence is estimated to be between 20,000 to 30,000 newly diagnosed patients each year in the US.

Core decompression of the hip is a minimally invasive surgical technique performed to manage symptoms in early stages (precollapse) of the condition. The procedure involves drilling holes into the femoral head to relieve pressure and create channels for new blood vessels to nourish the affected areas. Multiple adjuncts to core decompression, such as structural bone grafts, bone marrow concentrates, and bone proteins have been developed to accelerate the healing process in these patients. In recent years, considerable research activity has also been expanded to find new bone substitutes with osteoconductive properties (where bone grows on a surface) for the use in the treatment of surgically created defects.

Genex® Bone Graft Substitute is a catalyst for bone healing. It complements the body's natural healing processes and encourages normal bone structure to be restored at a steady rate. Over 12 months, the graft matrix is completely absorbed and replaced by bone. No foreign artifacts are left behind to impair structural integrity.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years or older with osteonecrosis of the femoral head
* Surgeon considers the patient appropriate for the core decompression procedure of the hip
* Subject provides voluntarily signature on the IRB approved Informed Consent Form
* Subject must be physically and mentally willing and able, in the Investigator's opinion at the time of enrollment, to be compliant with the protocol and complete the study protocol and follow ups

Exclusion Criteria:

* Subject is pregnant at the time of surgery
* Subject is incarcerated
* Subject is not comfortable with speaking, reading and understanding questions and providing responses in an available language for the questionnaires provided for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are 18 years or older with early osteonecrosis of the femoral head and meet the inclusion and exclusion criteria based on the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline X-ray result. | 6 weeks, 12 weeks, 6 months, 12 months post operatively
  Assessment of bone regeneration
Change from baseline MRI result. | 12 months
  Assessment for no further collapse or progression of osteonecrosis

SECONDARY OUTCOMES:
Numeric Pain Scale | Baseline, 6 weeks, 12 weeks, 6 months, 12 months
  To assess pain using the Numeric Pain Scale on a scale of 0-10 with 10 being the worst possible pain report and 0 being no pain
Modified Harris Hip Score | Baseline, 6 weeks, 12 weeks, 6 months, 12 months
  To evaluate the success of the core decompression procedure using the Modified Harris Hip Score by adding up the assigned points for each question, divided by a maximum score of (91) x 100 to create a percentage. A higher score equals a higher level of physical function (100% = full function).
Hip Outcome Score | Baseline, 6 weeks, 12 weeks, 6 months, 12 months
  To assess the outcome of the treatment intervention using the Hip Outcome Score with five possible responses, graded from 0 to 4 with 4 being no difficulty at all and 0 unable to do in regard to physical limitations.
EQ-5D-5L Score | Baseline, 6 weeks, 12 weeks, 6 months, 12 months
  To assess aspects of mobility, self-care, usual activities, pain/discomfort and anxiety/depression using the EQ-5D-5L tool. The EQ-5D-5L descriptive system uses (1) 'not /no problems', (2) 'slight problems', (3) 'moderate problems', (4) 'severe problems', and (5) 'unable to' (mobility, self-care, usual activities), 'extreme' (pain/depression), or 'extremely' (anxiety/depression).

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Piuzzi, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moya-Angeler J, Gianakos AL, Villa JC, Ni A, Lane JM. Current concepts on osteonecrosis of the femoral head. World J Orthop. 2015 Sep 18;6(8):590-601. doi: 10.5312/wjo.v6.i8.590. eCollection 2015 Sep 18. PMID 26396935
- [Background] Weinstein RS. Glucocorticoid-induced osteonecrosis. Endocrine. 2012 Apr;41(2):183-90. doi: 10.1007/s12020-011-9580-0. Epub 2011 Dec 15. PMID 22169965
- [Background] Yang HL, Zhu XS, Chen L, Chen CM, Mangham DC, Coulton LA, Aiken SS. Bone healing response to a synthetic calcium sulfate/beta-tricalcium phosphate graft material in a sheep vertebral body defect model. J Biomed Mater Res B Appl Biomater. 2012 Oct;100(7):1911-21. doi: 10.1002/jbm.b.32758. Epub 2012 Jul 30. PMID 22847979